CLINICAL TRIAL: NCT05736627
Title: Learning Effect of Onsite vs. Online Education in a Medical Context
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Copenhagen Academy for Medical Education and Simulation (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Hanne Tonnesen, Professor, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Online learning effect
Record Dates: First submitted 2023-02-01; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Online Learning
MeSH Terms: interventions — Pharmaceutical Services, Online

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The randomisation result will be opened for course participants and investigator when sending out the welcome letter about 3 weeks prior to running the course.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online setting (Experimental): Research course delivered digitally (Zoom or Teams meeting rooms) at a distance.
  Interventions: Other: Online
- Onsite setting (No Intervention): Research course delivered physically in educational facilities.

INTERVENTIONS:
Other: Online — Online research course delivered live digitally at a distance.
  Arms: Online setting

SUMMARY:
The goal of this clinical trial is to learn about the effects of online medical education in PhD students. The main question it aims to answer is:

What is the effect of onsite compared to online research courses on theoretical knowledge of research methodology and motivation for young medical researchers? Participants will join 20 research courses which are computer randomised to be delivered online (intervention) or onsite (control group) with 10-12 PhD students of each course (200-240 participants). Participants will be followed for up to two years after their course. The outcomes are

* theoretical learning (main)
* academic achievements
* motivation
* self-efficacy

Researchers will compare online and onsite research courses to see if there is a difference in theoretical learning, academic achievements, motivation and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* All PhD students on the courses if they are able to give informed consent

Exclusion Criteria:

* Declining to participate
* Withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Theoretical learning | Up to 3 months
  "Knows" or "Knows how" according to Miller's Pyramid of Competence measured by MCQ

SECONDARY OUTCOMES:
Academic achievement | Up to 25 months
  Measured by Google Scholar Profile (number of publications, number of citations, H-index and i10-index
Motivation | Up to 3 months
  Intrinsic Motivation Inventory
Self-efficacy | Up to 3 months
  Williams and Smith's single item measure of self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Rie Raffing, Frederiksberg, Frederiksberg Hospital, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raffing R, Konge L, Tonnesen H. Learning effect of online versus onsite education in health and medical scholarship - protocol for a cluster randomized trial. BMC Med Educ. 2024 Aug 26;24(1):927. doi: 10.1186/s12909-024-05915-z. PMID 39187817